CLINICAL TRIAL: NCT04719975
Title: The Electrophysiological Signature of the Mental Fatigue-induced Impairment in Endurance Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MF-EEG-MRCP
Record Dates: First submitted 2020-09-22; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Mental Fatigue; Electroencephalography
MeSH Terms: conditions — Mental Fatigue | interventions — Stroop Test

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, counter-balanced, cross-over design
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mental Fatigue (Stroop) - Chair task (Experimental): Participants will be performing the Chair Task (150 submaximal dynamic knee extensions at 50% of their maximal voluntary contraction (MVC)) when mentally fatigued. A 60 minute variant of the Stroop task will be used to induce the mental fatigue. During the whole trial EEG will be measured.
  Interventions: Other: Mental Fatigue (Stroop task)
- Control Task (Documentary) - Chair Task (Placebo Comparator): In the control task subjects will have to watch a documentary on the same computer screen as that used for the experimental trial. These documentaries are chosen based on their emotionally neutral, yet engaging content. This will be followed by the Chair Task, During the whole trial EEG will be measured.
  Interventions: Other: Control (Documentary)
- Mental Fatigue (Stroop) - Bike Task (Experimental): Participants will be performing the Bike Task (a 9 min cycling task performed at 45 rpm with intensity being constant and will be 10% below VT) when mentally fatigued. A 60 minute variant of the Stroop task will be used to induce the mental fatigue. During the whole trial EEG will be measured.
  Interventions: Other: Mental Fatigue (Stroop task)
- Control task (Documentary) - Bike Task (Placebo Comparator): In the control task subjects will have to watch a documentary on the same computer screen as that used for the experimental trial. These documentaries are chosen based on their emotionally neutral, yet engaging content. This will be followed by the Bike Task, During the whole trial EEG will be measured.
  Interventions: Other: Control (Documentary)

INTERVENTIONS:
Other: Mental Fatigue (Stroop task) — A modified Stroop task of approximately 60 min will be used in order to induce mental fatigue (MF). This will be based on their performance during the max test that was conducted during the familiarization session. In this task, which will be partitioned in 4 blocks of 468 stimuli, four colored words ("rood", "blauw", "groen" and "geel") will be presented one at a time on a computer screen. The participants will be required to indicate the color of the word, ignoring the meaning of the word itself.
  Arms: Mental Fatigue (Stroop) - Bike Task; Mental Fatigue (Stroop) - Chair task
Other: Control (Documentary) — In the control task subjects will have to watch a documentary of 60 min on the same computer screen as the one used for the experimental trial. In order to avoid under- and over-arousal the subjects will have the opportunity to choose between several documentaries as proposed by the research team. During the control task physiological and psychological measures will be assessed at the same time points as during the mental fatigue trial.
  Arms: Control Task (Documentary) - Chair Task; Control task (Documentary) - Bike Task

SUMMARY:
The purpose of this project is to provide further insights into the neurophysiology behind the MF-induced impairment in endurance performance. The aim is to perform a randomized controlled trial in which we partly replicate studies of Marcora et al. (2009) and Bigliassi et al. (2017), while extensively monitoring brain activity during the entire protocol (i.e. both cognitive and physical tasks) by using EEG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological or cardiovascular disorders)
* Male or female
* No medication
* Non-smoker
* Between 18 and 35 years old
* Recreational athlete population (performance level 2 or 3 for men according to De Pauw et al. (2013) and performance level 2 or 3 for woman according to Decroix et al. (2016)

Exclusion Criteria:

* Injuries over the last 6 months
* Suffering from any cardiovascular condition
* Use of medication
* Suffering from other health conditions at the time of testing
* Use of caffeine or alcohol 24 hours prior to each trial
* Heavy efforts 24 hours prior to each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram data | 1 hours 30 minutes - 2 hours
  During whole of the trials EEG data will be gathered, each trial will last one and a half to two hours. EEG power in delta, theta, alpha, beta band.
Reaction Time Flanker Task | Total of 10 minutes
  Reaction Time will be assessed during Flanker task
Accuracy Flanker Task | Total of 10 minutes
  Accuracy will be assessed during Flanker task
Reaction Time Stroop Task | 60 minutes
  Reaction Time will be assessed during Stroop task
Accuracy performance Stroop Task | 60 minutes
  Accuracy will be assessed during Stroop task

CONTACTS AND LOCATIONS:
Locations (1):
- Human Physiology and Sports Physiotherapy Research Group, Brussels, Elsene, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proost M, Habay J, DE Wachter J, DE Pauw K, Marusic U, Meeusen R, DE Bock S, Roelands B, VAN Cutsem J. The Impact of Mental Fatigue on a Strength Endurance Task: Is There a Role for the Movement-Related Cortical Potential? Med Sci Sports Exerc. 2024 Mar 1;56(3):435-445. doi: 10.1249/MSS.0000000000003322. Epub 2023 Oct 16. PMID 37847068